CLINICAL TRIAL: NCT02285842
Title: Post Market Clinical Follow-Up Study Protocol for CONSERVE® Press-Fit Femoral Components
Status: Active, not recruiting | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-LJH-002F
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-04

CONDITIONS: Joint Disease
Keywords: osteoarthritis; avascular necrosis; ankylosis; protrusio acetabuli; painful hip dysplasia; rheumatoid arthritis; correction of functional deformity; revision procedures
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Osteonecrosis; Ankylosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary Hip Resurfacings: Single study group previously implanted with CONSERVE® Press-Fit Femoral Components
  Interventions: Device: Primary hip resurfacing device

INTERVENTIONS:
Device: Primary hip resurfacing device — CONSERVE® Press-Fit Femoral Components

SUMMARY:
MicroPort Orthopedics (MPO) is conducting this PMCF study to evaluate the safety and efficacy of its THA and resurfacing components marketed in the EU. These types of studies are required by regulatory authorities for all THA and resurfacing devices that do not have medium to long-term clinical evidence available at the time of gaining approval to market in the EU. This study has been designed in accordance with MEDDEV 2.12/2 rev 2.

DETAILED DESCRIPTION:
MicroPort Orthopedics Inc. (MPO) currently markets several total hip arthroplasty (THA) and resurfacing components throughout the world, including the European Union (EU). As part of the process for gaining approval to market in the EU, MPO is conducting this post market clinical follow-up (PMCF) study to evaluate the safety and efficacy of these components. The objectives of this study are to evaluate component survivorship, total functional outcome scores, and radiographic outcomes of implanted subjects at out to 10 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Has undergone primary hip resurfacing for any of the following:
* Non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis, ankylosis, protrusio acetabuli, or painful hip dysplasia;
* Inflammatory degenerative joint disease such as rheumatoid arthritis; or
* Correction of functional deformity
* Subject is implanted with the specified combination of components
* Subject is willing and able to complete required study visits or assessments

Exclusion Criteria:

* Subjects skeletally immature (less than 21 years of age) at time of primary resurfacing surgery
* Subjects currently enrolled in another clinical study which could affect the endpoints of this protocol
* Subjects unwilling to sign the Informed Consent document
* Subjects with substance abuse issues
* Subjects who are incarcerated or have pending incarceration

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been previously implanted with CONSERVE® Press-Fit Femoral Components
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Component Survivorship | 10 years post-operative
  The primary objective of this study is to estimate survivorship of all components at specified intervals out to 10 years follow-up.

SECONDARY OUTCOMES:
Patient functional outcomes | Screening (First Available), 2-5 years, 5-7 years, and 10 years
  To characterize total functional scores, as assessed by HOOS and EQ-5D-3L scores
Component alignment | Screening (First Available), 2-5 years, 5-7 years, and 10 years
  To evaluate component alignment (neck shaft angle, stem shaft angle, and cup inclination) and the presence of radiolucencies surrounding implanted components

CONTACTS AND LOCATIONS:
Overall Officials: Paul Beaule, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada